CLINICAL TRIAL: NCT02049060
Title: Phase I-Ib Study of the Combination of Tivantinib Plus Pemetrexed and Carboplatin as First-line Therapy in Patients With Advanced or Metastatic Cancer Suitable for a Carboplatin and Pemetrexed Regimen as Part of Their Specific Therapy
Brief Title: Study of the Combination of Tivantinib Plus Pemetrexed and Carboplatin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Principal Investigators, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2011-001
Record Dates: First submitted 2013-05-24; First posted 2014-01-29 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Malignant Pleural Mesothelioma; Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: MPM; NSCLC
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tivantinib+carboplatino+pemetrexed (Experimental): •- 1 level: Tivantinib 120 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  •0 level: Tivantinib 240 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  •+ 1 level: Tivantinib 360 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  Interventions: Drug: Tivantinib

INTERVENTIONS:
Drug: Tivantinib — •- 1 level: Tivantinib 120 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  •0 level: Tivantinib 240 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  •+ 1 level: Tivantinib 360 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks
  Other Names: ARQ 197

SUMMARY:
This is a prospective, open-label, mono-centric, phase I-Ib trial of Tivantinib in combination with Pemetrexed and Carboplatin as first-line therapy in patients with advanced or metastatic cancer suitable for a Carboplatin and Pemetrexed regimen as part of their specific therapy.

DETAILED DESCRIPTION:
This is a prospective, open-label, mono-centric, phase I-Ib trial of Tivantinib in combination with Pemetrexed and Carboplatin as first-line therapy in patients with advanced or metastatic cancer suitable for a Carboplatin and Pemetrexed regimen as part of their specific therapy.This trial will be conducted to determine the maximum tolerated dose (MTD), safety/tolerability, pharmacokinetics and preliminary anti-tumor activity of escalating doses of Tivantinib in combination with standard fixed doses of Carboplatin and Pemetrexed.

The dose-escalation stage will be followed by an expansion stage at the MTD to better define toxicity and clinical activity. MTD is defined as the highest dose level at which < 33% of 6 patients experience a DLT.

Eligible patients will be enrolled and treated according to the following 3 + 3 design starting from cohort 0:

* 1 level: Tivantinib 120 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks 0 level: Tivantinib 240 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks

  * 1 level: Tivantinib 360 mg p.o. BID + Carboplatin AUC 5 i.v. day 1 every 3 weeks + Pemetrexed 500 mg/mq i.v. day 1 every 3 weeks

If the frequency of DLTs encountered at dose-level +1 will not fulfil the MTD definition, then Tivantinib 360 mg bid in combination with Carboplatin AUC 5 and Pemetrexed 500 mg/mq will be accepted as the recommended dose for phase IItrials.

Treatment will be continued on the basis of tumor assessment. Patients with stable disease, complete or partial response will continue treatment until progressive disease, unacceptable toxicity, patient or physician decision. For chemotherapy agents, however, a maximum of 6 cycles will be administered. Tivantinib will be continued until progressive disease, unacceptable toxicity, patient or physician decision.

Toxicity will be graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.

Following the dose-escalation phase of the study, additional patients (in order to reach a total of 13 patients with MPM and 18 patients with NSCLC treated at MTD/recommended dose for phase Ib trials) will be accrued to the expansion stage of this trial, to assess the preliminary anti-tumor activity of Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq) primarily.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with MPM or non squamous NSCLC.
2. Inoperable disease according to local surgeon, not previously treated with chemotherapy; patients relapsed/progressed after previous surgery will be also evaluable for inclusion.
3. Age > 18.
4. ECOG Performance Status 0-1 and life expectancy of at least 12 weeks.
5. Measurable and/or evaluable lesions according to modified RECIST criteria [51].
6. Written informed consent.
7. Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating center.
8. Patients must use effective contraception during the study lasting at least one month after the end of treatment for both sexes.
9. Laboratory requirements:

   * Neutrophils >1.5 x 109/L and Platelets >100 x 109/L
   * Total bilirubin <1.5 time the upper-normal limits (UNL) of the Institutional normal values, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, or <5 x UNL in case of liver metastases, alkaline phosphatase <2.5 x UNL, < 5 x UNL in case of liver metastases, <10 x UNL in case of bone metastases.
   * Creatinine clearance >50 mL/min

Exclusion Criteria:

1. Any prior chemotherapy (including intracavitary administration).
2. Symptomatic and/or unstable pre-existing brain metastases.To be enrolled in the study , subjects must have confirmation of stable disease by MRI or computer tomography (CT) scan within 4 weeks from day 1 of cycle 1 of treatment and have CNS metastases well controlled by steroids, anti - epileptics or other symptom-relieving medications
3. Serious non-healing wound or ulcer.
4. Evidence of bleeding diathesis or coagulopathy.
5. Uncontrolled hypertension.
6. Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents (<6 months), myocardial infarction (< 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
7. Current treatment with anticoagulants for therapeutic purposes.
8. Treatment with any investigational drug within 30 days prior to enrolment.
9. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
11. Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities (DLTs) of Tivantinib | 18 months
  1.To determine the dose limiting toxicities (DLTs) of Tivantinib given orally twice daily on a continuous schedule in combination with Carboplatin and Pemetrexed administered intra-venous every 3 weeks.

SECONDARY OUTCOMES:
To determine the pharmacokinetics profile of Tivantinib in combination with Carboplatin and Pemetrexed | 18 months
  To determine the pharmacokinetics profile of Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq).
To assess the preliminary anti-tumor activity of Tivantinib with PFS | 18 months
  To assess the preliminary anti-tumor activity of Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq), in terms of 3-months progression-free survival rate for malignant pleural mesothelioma patients and 5-months progression-free survival rate for NSCLC patients
To assess the preliminary anti-tumor activity of Tivantinib with RECIST | 18 months
  To assess the preliminary anti-tumor activity of Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq), in terms of objective response rate according to "response criteria evaluation criteria in solid tumors" (Modified RECIST criteria for Malignant Pleural Mesothelioma), and duration of response.
To evaluate dynamic changes in blood levels | 18 months
  To evaluate dynamic changes in blood levels of hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), and soluble c-Met, in patients treated with Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq)
To evaluate the expression of biomarkers | 18 months
  To evaluate the expression of phospho-c-Met, total c-Met, and downstream markers of c-Met signaling pathway in patients' tumor tissue samples
To dermine the MTD of combination | 18 month
  To determine the MTD of the combination, defined as the highest dosage cohort at which no more than one of six patients experiences a DLT during the first treatment cycle, considering the level +1 as the maximum level to explore. This will be the recommended dose for a subsequent phase II study.
To assess the preliminary anti-tumor activity of tivantinib | 18 month
  To assess the preliminary anti-tumor activity of Tivantinib in combination with Carboplatin (AUC 5) and Pemetrexed (500 mg/mq), in terms of 3-months progression-free survival rate for malignant pleural mesothelioma patients and 5-months progression-free survival rate for NSCLC patients

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
not planned